CLINICAL TRIAL: NCT01138449
Title: Efficacy of Neonatal Vitamin A Supplementation in Improving Child Survival in Haryana, India: Generation of Evidence Necessary for Informing Global Policy
Brief Title: Efficacy of Newborn Vitamin A Supplementation Versus Placebo in Improving Child Survival (NeoVitA Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, NBhandari, Director, Society for Applied Studies
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RPC356; UTRN 112336978-06032010834860 (Registry Identifier: Clinical Trial Registry-India)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Neonatal Vitamin A Supplementation
Keywords: Vitamin A; Neonatal mortality; Infant mortality
MeSH Terms: conditions — Infant Death | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin A (Experimental): Vitamin A capsules have retinol palmitate (50,000 IU) and minute amounts of vitamin E in soybean oil
  Interventions: Drug: Vitamin A
- Placebo (Placebo Comparator): Placebo capsules contain minute amounts of vitamin E in soybean oil
  Interventions: Drug: Vitamin A

INTERVENTIONS:
Drug: Vitamin A — Retinol palmitate (50,000 IU) and minute amounts of vitamin E in soybean oil, orally as a single dose to neonates on the day of birth or in the next 2 days of birth keeping a minimum period of 2 hours between the birth and the dosing

SUMMARY:
The study is a large randomized controlled trial to assess the efficacy and safety of neonatal vitamin A supplementation administered to neonates once orally either on the day of birth or in the next 2 days in improving infant survival in the first 6 months of life.

DETAILED DESCRIPTION:
The study is an individually randomized trial conducted in two districts in the state of Haryana.

Community informants report births to the enrolment team. At enrolment, the team explains the study to the family and in those willing, written consent is obtained from the parents of the infant. The infant is given the dose of vitamin A/placebo and a form containing baseline socioeconomic characteristics and information on feeding practices of the infant and mother is filled.

After enrollment, each infant is visited by the enrollment team at hospital or home 1 day and 3 days after supplementation to document any illnesses in the baby. Newborns with illnesses are referred/escorted to the nearest health facility for management.

Enrolled infants are visited when aged 29 days, 3, 6 and 12 months to document vital status and hospitalizations since the last visit. Information on feeding practices, immunization, maternal intake of vitamin A rich foods and supplements, and intake of any supplement containing vitamin A by the infant is recorded at these visits. Subgroup analyses includes the effect of vitamin A supplementation in LBW and non LBW infants, male and female infants, immunized and unimmunized infants, infants of families in the poorest and richest quintiles and by vitamin A intake of mothers. For all deaths, verbal autopsy interviews are conducted.

Blood specimens are obtained in a subsample of infants at 2 weeks and 3 months of age and in a subsample of mothers at 3 months of age.

Quality control activities include independent and supervised checks and are conducted for a subsample by a separate team.

A DSMB has been constituted for the study. All deaths occurring within 72 hours of supplementation will be reported to the SAS ERC and to the WHO Coordinating Unit.

At the recent DSMB meeting in February 2012, the DSMB recommended an increase in sample size to 45,000 instead of the earlier estimate of 40,200 because of somewhat lower than expected mortality rates. This increase in sample size is expected to preserve the specified power of 0.85 and the corresponding level of precision anticipated at the design stage.

Similar trials are being funded by the World Health Organization (Geneva) in Ghana and Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate
* All births in the study area that are contacted by enrolment team within the eligible age window

Exclusion Criteria:

* Unable to feed on offering feeds, as reported by the mother
* Mother does not intend to stay in the study area for at least 6 months

Ages: 2 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44984 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Risk of death | Period between receiving the intervention/placebo and six months of age
  To determine if vitamin A supplementation (50,000 IU) given to neonates once orally either on the day of birth or in the next 2 days will reduce mortality in the first half of infancy as compared to placebo.

SECONDARY OUTCOMES:
Risk of death | Period between receiving the intervention/placebo and 28 days of age
  To determine the efficacy of vitamin A supplementation (50,000 IU) given to neonates once orally either on the day of birth or in the next 2 days in reducing mortality in the neonatal period (first month of life).
Risk of death | Period between receiving the intervention/placebo and 12 months of age
  To determine the efficacy of vitamin A supplementation (50,000 IU) given to neonates once orally either on the day of birth or in the next 2 days in reducing mortality at 12 months.
Risk of hospital admission | Period between receiving the intervention/placebo and six months of age
  To determine the efficacy of the above intervention in reducing the incidence of severe morbidity defined as hospitalizations due to any illness in the first 6 months of infancy.
Bulging fontanelle, vomiting, irritability, fever, diarrhea, inability to suck or feed, convulsions or any other conditions that caused parents to be concerned | Three day period following supplementation
  To assess bulging fontanelle, vomiting, irritability, fever, diarrhea, inability to suck or feed, convulsions or any other conditions that caused parents to be concerned, in the 3 day period following administration of the supplement
Vitamin A status in a subgroup of newborns and caregivers in the intervention and placebo groups | Two weeks and three months of age
  To determine vitamin A status in a subsample of infants and caregivers in the intervention and placebo groups at 2 weeks and 3 months of age in the vitamin A supplementation and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, MD, PhD, Principal Investigator — Society for Applied Studies; Sunita Taneja, MD, PhD, Principal Investigator — Society for Applied Studies; Sarmila Mazumder, MD, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] NEOVITA Study Author Group; Bahl R, Bhandari N, Dube B, Edmond K, Fawzi W, Fontaine O, Kaur J, Kirkwood BR, Martines J, Masanja H, Mazumder S, Msham S, Newton S, Oleary M, Ruben J, Shannon C, Smith E, Taneja S, Yoshida S. Efficacy of early neonatal vitamin A supplementation in reducing mortality during infancy in Ghana, India and Tanzania: study protocol for a randomized controlled trial. Trials. 2012 Feb 23;13:22. doi: 10.1186/1745-6215-13-22. PMID 22361251
- [Result] Mazumder S, Taneja S, Bhatia K, Yoshida S, Kaur J, Dube B, Toteja GS, Bahl R, Fontaine O, Martines J, Bhandari N; Neovita India Study Group. Efficacy of early neonatal supplementation with vitamin A to reduce mortality in infancy in Haryana, India (Neovita): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Apr 4;385(9975):1333-42. doi: 10.1016/S0140-6736(14)60891-6. Epub 2014 Dec 11. PMID 25499546
- [Derived] Upadhyay RP, Martines JC, Taneja S, Mazumder S, Bahl R, Bhandari N, Dalpath S, Bhan MK. Risk of postneonatal mortality, hospitalisation and suboptimal breast feeding practices in low birthweight infants from rural Haryana, India: findings from a secondary data analysis. BMJ Open. 2018 Jun 22;8(6):e020384. doi: 10.1136/bmjopen-2017-020384. PMID 29934384